CLINICAL TRIAL: NCT04576143
Title: Efficacy and Safety of Dose-dense Epirubicin and Cyclophosphamide Plus Paclitaxel as Neoadjuvant Chemotherapy for HER2-negative Early Breast Cancer：a Multicenter Randomized Controlled Trial
Brief Title: Efficacy and Safety of Dose-dense Chemotherapy (ddEC-ddP) for Neoadjuvant Chemotherapy of HER2-negative Breast Cancer
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Women's Hospital School Of Medicine Zhejiang University (Other); Changxing People's Hospital (Other); Zhejiang Provincial People's Hospital (Other); Hangzhou First People's Hospital, School of Medicine, Zhejiang Universiry (Unknown); Huizhou Municipal Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-495
Record Dates: First submitted 2020-09-20; First posted 2020-10-06 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-01

CONDITIONS: HER2-negative Breast Cancer; Neoadjuvant Chemotherapy
Keywords: HER2-negative breast cancer; dose-dense chemotherapy; preoperative neoadjuvant chemotherapy; EC-T; ddEC-ddP
MeSH Terms: interventions — Epirubicin; Cyclophosphamide; Docetaxel; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- epirubicin/CTX × 4 - docetaxel × 4, every 3 weeks a cycle (Active Comparator): Cycle 1-4: Epirubicin i.v. 90 mg/m2, Cyclophosphamide i.v. 600 mg/m2 (One cycle = 21 days); Cycle 5-8: Docetaxel i.v. 100mg/m2 (One cycle = 21 days) .
  Interventions: Drug: Epirubicin; Drug: Cyclophosphamid; Drug: Docetaxel
- epirubicin/CTX × 4 - paclitaxel × 4, every 2 weeks a cycle (Experimental): Cycle 1-4: Epirubicin i.v. 90 mg/m2, Cyclophosphamide i.v. 600 mg/m2 (One cycle = 14 days); Cycle 5-8:Paclitaxel i.v. 175mg/m2 (One cycle = 14 days) .
  Interventions: Drug: Epirubicin; Drug: Cyclophosphamid; Drug: Paclitaxel

INTERVENTIONS:
Drug: Epirubicin — i.v. 90 mg/m2
  Other Names: Epirubicin Hydrochloride
Drug: Cyclophosphamid — i.v. 600 mg/m2
  Other Names: CTX
Drug: Docetaxel — i.v. 100 mg/m2
  Arms: epirubicin/CTX × 4 - docetaxel × 4, every 3 weeks a cycle
Drug: Paclitaxel — i.v. 175 mg/m2
  Other Names: PTX
  Arms: epirubicin/CTX × 4 - paclitaxel × 4, every 2 weeks a cycle

SUMMARY:
Recent clinical studies showed that breast cancer patients especially for those with lymph node metastasis may benefit from dose-dense chemotherapy, like adriamycin and cyclophosphamide (AC) q2w×4→ paclitaxel (P) q2w×4. However, the studies on dose-dense (dd) regimen chemotherapy is mostly based on postoperative adjuvant chemotherapy and the optimum of dose-dense chemotherapy has not been determined for Chinese population with HER2-negative breast cancer patients. In our study, a prospective, randomized, open-label, multi-center clinical study was conducted to compare the efficacy and safety of dose-dense chemotherapy regimen (dd epirubicin/cyclophosphamide (EC) followed by dd paclitaxel (P)) and conventional chemotherapy (epirubicin/cyclophosphamide (EC) followed by docetaxel (T)) as preoperative neoadjuvant chemotherapy in the treatment of HER2-negative breast cancer in Chinese population.

DETAILED DESCRIPTION:
Neoadjuvant chemotherapy refers to systemic chemotherapy as the first step for treating breast cancer patients before planned local treatment like surgery for those without distant metastasis. Randomized trials of chemotherapy have demonstrated similar long-term outcomes when patients were given the same treatment preoperatively compared with postoperatively. It is reported that preoperative neoadjuvant chemotherapy can facilitate breast conservation, render inoperable tumors operable and provide important prognostic information at an individual patient level based on response to therapy.

According to the recommendation of National Comprehensive Cancer Network (NCCN) guideline, patients with inoperable breast cancer, such as inflammatory breast cancer, N3 nodal disease and T4 tumors are candidates for preoperative systemic therapy. As for those operable patients with HER2-positive disease and triple-negative breast cancer (TNBC), if T ≥2 or N ≥1, or large primary tumor relative to breast size in a patient who desires breast conservation, neoadjuvant chemotherapy is also preferred. Based on the results of NSABP-27 and Aberdeen clinical trials, chemotherapeutic drugs including taxanes (such as docetaxel, paclitaxel) and anthracyclines (such as doxorubicin, epirubicin) have become the standard neoadjuvant chemotherapy regimens for early operable patients and for HER2-negative breast cancer patients, anthracyclines combined with cyclophosphamide followed by docetaxel is mostly common used.

Limited to myelosuppression and bone marrow repair, conventional chemotherapy cycle is usually set once every 3-4 weeks. Recent years, the application of granulocyte colony stimulating factor (G-CSF), which can shorten the recovery time of leukocytes, enables dose-dense chemotherapy (maximum tolerable dose, every 2 weeks as a cycle) to become a treatment option for high-risk patients. The concept of dose-dense chemotherapy is based on a mathematical model developed by Norton and Simon, and relies on an understanding of Gompertzian model of tumor growth. Gompertzian kinetics explain that human neoplasms do not grow in an exponential fashion, instead the cell-doubling time becomes progressively longer as the tumor growth. Thus, cancer treatments that reduce the size of a tumor can promote faster tumor regrowth between treatments indirectly. So Norton-Simon hypothesis suggests that the most effective strategy is to expose the tumor to cytotoxic agents as frequently as possible to minimize regrowth between cycles.

The CALGB 9471 used a randomized, 2×2 factorial design to prospectively compare sequential doxorubicin, paclitaxel, cyclophosphamide with concurrent doxorubicin and cyclophosphamide followed by paclitaxel, and to compare dose-dense schedules with conventional schedules. A total of 2005 node-positive, previously untreated patients were enrolled. At a median follow-up of 36 months, dose-dense treatment significantly improved disease-free survival (DFS) and overall survival (OS) compared with conventionally scheduled treatment. The GIM2 study also demonstrated that dose-dense adjuvant chemotherapy (FEC-P and EC-P every 2 weeks a cycle) improved DFS and OS compared with standard interval chemotherapy (every 3 weeks a cycle). However, the studies on dose-dense chemotherapy is mostly based on postoperative adjuvant chemotherapy. We aim to conduct a prospective, randomized, open-label, multi-center clinical study to compare the efficacy and safety of dose-dense chemotherapy (dd epirubicin/cyclophosphamide (EC) followed by dd paclitaxel (P)) and conventional chemotherapy (epirubicin/cyclophosphamide (EC) followed by docetaxel (T)) as preoperative neoadjuvant chemotherapy in the treatment of HER2-negative breast cancer in Chinese population.

ELIGIBILITY:
Inclusion Criteria:

1. Female aged 18-70 years old;
2. Histological confirmed with unilateral invasive carcinoma (all pathological types are applicable), clinical stage IIA-IIIA;
3. Definite reports on ER/PR/HER2 receptor showing all HER2 negative (HER2 is 0~1+ or 2+ but determined negative via fluorescence in situ hybridization (FISH) or chemiluminescent in situ hybridization (CISH) detected (no amplification) is defined as HER2 negative);
4. According to RECIST 1.1, there is at least one measurable objective focus, tumor size > 2cm;
5. Eastern Cooperative Oncology Group (ECOG) performance score is 0 or 1;
6. Cardiac function: left ventricular ejection fraction (LVEF)≥55%;
7. Normal bone marrow function: White blood cell count > 4 × 10^9/l, neutrophil count > 1.5 × 10^9/l, platelet count > 100 × 10^9/l and hemoglobin 9g/dl;
8. Normal liver and renal function: aspartate aminotransferase (AST) and ALT ≤2.5 folds of the upper limit of normal values, total bilirubin ≤1.5 folds of the upper limit of normal values; Serum creatinine ≤1.5 folds of the upper limit of normal value.
9. Informed consent form signed.

Exclusion Criteria:

1. HER2 is positive;
2. Metastasis at any location;
3. Previous neoadjuvant therapy, including chemotherapy, radiotherapy and hormone therapy;
4. Severe systemic disease and/or uncontrollable infection, unable to be enrolled in this study;
5. Known allergic or intolerable to chemotherapeutic agents;
6. Previously suffering from malignant tumors within 5 years (except for basal cell carcinoma and cervical carcinoma in situ), including contralateral breast cancer;
7. Cardiovascular disease: LVEF <50% (echocardiography) of New York Heart Association (NYHA) ≥ grade 2;
8. Pregnant and breast-feeding women; Pregnancy test showed positive results before drug administration after enrolling in to the study; Women at childbearing age refuse to take contraception measures during the treatment and 8 weeks after completion of treatment;
9. Already enrolled into other clinical trials;
10. The researchers judged the patients who were not suitable for this study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2020-09-20 (Actual); Primary Completion 2023-06-20 (Estimated); Study Completion 2027-09-20 (Estimated)

PRIMARY OUTCOMES:
pathological complete response (pCR) | Following the completion of 16 weeks or 24 weeks of neoadjuvant chemotherapy Treatment.
  pCR is defined as the absence of noninvasive tumor residuals in breast and axillary lymph nodes (ypT0/is ypN0) after neoadjuvant therapy.

SECONDARY OUTCOMES:
objective response rate (ORR) | Following the completion of 16 weeks or 24 weeks of neoadjuvant chemotherapy Treatment.
  ORR is defined as the proportion of patients who achieved a complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST).
disease free survival (DFS) | Time of Surgery up to 5 years
  Events including local relapse, distant metastasis, contralateral breast cancer, second primary cancer or death from any cause
breast-conserving rate (BCR) | Following the completion of 16 weeks or 24 weeks of neoadjuvant chemotherapy Treatment.
  The rate of patients who were performed breast-conserving surgery.
Number of participants with adverse events | First Dose of chemotherapy up to 12 months.
  (like cardiotoxicity ,hematological toxicity，gastrointestinal symptoms) as a measure of safety

CONTACTS AND LOCATIONS:
Overall Officials: Yiding Chen, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wolmark N, Wang J, Mamounas E, Bryant J, Fisher B. Preoperative chemotherapy in patients with operable breast cancer: nine-year results from National Surgical Adjuvant Breast and Bowel Project B-18. J Natl Cancer Inst Monogr. 2001;(30):96-102. doi: 10.1093/oxfordjournals.jncimonographs.a003469. PMID 11773300
- [Background] Rastogi P, Anderson SJ, Bear HD, Geyer CE, Kahlenberg MS, Robidoux A, Margolese RG, Hoehn JL, Vogel VG, Dakhil SR, Tamkus D, King KM, Pajon ER, Wright MJ, Robert J, Paik S, Mamounas EP, Wolmark N. Preoperative chemotherapy: updates of National Surgical Adjuvant Breast and Bowel Project Protocols B-18 and B-27. J Clin Oncol. 2008 Feb 10;26(5):778-85. doi: 10.1200/JCO.2007.15.0235. PMID 18258986
- [Background] Bear HD, Anderson S, Brown A, Smith R, Mamounas EP, Fisher B, Margolese R, Theoret H, Soran A, Wickerham DL, Wolmark N; National Surgical Adjuvant Breast and Bowel Project Protocol B-27. The effect on tumor response of adding sequential preoperative docetaxel to preoperative doxorubicin and cyclophosphamide: preliminary results from National Surgical Adjuvant Breast and Bowel Project Protocol B-27. J Clin Oncol. 2003 Nov 15;21(22):4165-74. doi: 10.1200/JCO.2003.12.005. Epub 2003 Oct 14. PMID 14559892
- [Background] Heys SD, Hutcheon AW, Sarkar TK, Ogston KN, Miller ID, Payne S, Smith I, Walker LG, Eremin O; Aberdeen Breast Group. Neoadjuvant docetaxel in breast cancer: 3-year survival results from the Aberdeen trial. Clin Breast Cancer. 2002 Oct;3 Suppl 2:S69-74. doi: 10.3816/cbc.2002.s.015. PMID 12435290
- [Background] Citron ML, Berry DA, Cirrincione C, Hudis C, Winer EP, Gradishar WJ, Davidson NE, Martino S, Livingston R, Ingle JN, Perez EA, Carpenter J, Hurd D, Holland JF, Smith BL, Sartor CI, Leung EH, Abrams J, Schilsky RL, Muss HB, Norton L. Randomized trial of dose-dense versus conventionally scheduled and sequential versus concurrent combination chemotherapy as postoperative adjuvant treatment of node-positive primary breast cancer: first report of Intergroup Trial C9741/Cancer and Leukemia Group B Trial 9741. J Clin Oncol. 2003 Apr 15;21(8):1431-9. doi: 10.1200/JCO.2003.09.081. Epub 2003 Feb 13. PMID 12668651
- [Background] Del Mastro L, De Placido S, Bruzzi P, De Laurentiis M, Boni C, Cavazzini G, Durando A, Turletti A, Nistico C, Valle E, Garrone O, Puglisi F, Montemurro F, Barni S, Ardizzoni A, Gamucci T, Colantuoni G, Giuliano M, Gravina A, Papaldo P, Bighin C, Bisagni G, Forestieri V, Cognetti F; Gruppo Italiano Mammella (GIM) investigators. Fluorouracil and dose-dense chemotherapy in adjuvant treatment of patients with early-stage breast cancer: an open-label, 2 x 2 factorial, randomised phase 3 trial. Lancet. 2015 May 9;385(9980):1863-72. doi: 10.1016/S0140-6736(14)62048-1. Epub 2015 Mar 2. PMID 25740286
- [Background] Earl HM, Hiller L, Dunn JA, Blenkinsop C, Grybowicz L, Vallier AL, Gounaris I, Abraham JE, Hughes-Davies L, McAdam K, Chan S, Ahmad R, Hickish T, Rea D, Caldas C, Bartlett JMS, Cameron DA, Provenzano E, Thomas J, Hayward RL; ARTemis Investigators Group. Disease-free and overall survival at 3.5 years for neoadjuvant bevacizumab added to docetaxel followed by fluorouracil, epirubicin and cyclophosphamide, for women with HER2 negative early breast cancer: ARTemis Trial. Ann Oncol. 2017 Aug 1;28(8):1817-1824. doi: 10.1093/annonc/mdx173. PMID 28459938